CLINICAL TRIAL: NCT07289581
Title: Effetto Del Trattamento Con Acido Butirrico Sull'Anoressia Nervosa
Brief Title: Effect of Treatment With Butyric Acid in Anorexia Nervosa
Acronym: AN-BUTIX
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 29252_spe; 29252 (Registry Identifier: Comitato Etico Area Vasta Centro - CEAVC)
Record Dates: First submitted 2025-12-01; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Anorexia Nervosa; Gut Microbiota; Weight Trajectory
Keywords: anorexia nervosa; gut microbiota; butyric acid; outcome
MeSH Terms: conditions — Anorexia Nervosa; Body-Weight Trajectory

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: Butyric Acid (Active Comparator): Participants with anorexia nervosa receiving butyric acid supplementation plus Treatment As Usual.
  Interventions: Dietary Supplement: Dietary Supplement: Butyric Acid
- Placebo Comparator: Placebo (Placebo Comparator): Participants with anorexia nervosa receiving placebo capsules plus Treatment As Usual.
  Interventions: Dietary Supplement: Dietary Supplement: Butyric Acid

INTERVENTIONS:
Dietary Supplement: Dietary Supplement: Butyric Acid — Daily oral supplementation with 2 capsules of microencapsulated butyric acid (Butyrose®, 550 mg each; total daily dose 1,100 mg) for 3 months, administered in addition to Treatment As Usual (nutritional rehabilitation + cognitive-behavioral therapy).
  Arms: Active Comparator: Butyric Acid
Dietary Supplement: Dietary Supplement: Butyric Acid — Daily oral supplementation with 2 placebo capsules matched in appearance and composition (maltodextrins, cellulose, inert excipients), administered for 3 months in addition to Treatment As Usual.
  Arms: Placebo Comparator: Placebo

SUMMARY:
This clinical trial aims to evaluate the therapeutic potential of oral butyric acid supplementation in individuals with anorexia nervosa (AN). T The study will assess whether butyric acid, administered alongside standard multidisciplinary care, improves weight restoration and contributes to overall clinical recovery.

The primary objectives are to determine:

- Whether butyric acid enhances weight restoration during the first 3 months of treatment.

Participants will be randomly assigned to receive either butyric acid or a placebo for 3 months, in addition to treatment-as-usual, which includes nutritional rehabilitation and cognitive-behavioral therapy.

Throughout the study, researchers will monitor:

* Changes in body weight and Body Mass Index (BMI)
* General and eating-disorder-related psychopathology
* Blood-based biomarkers related to inflammation, metabolism, and neuroendocrine function
* Gut microbiota composition and metabolites, including short-chain fatty acids

A total of 50 participants with AN are expected to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age 18-65 years
* Current diagnosis of Anorexia Nervosa (DSM-5)
* Able and willing to provide informed consent
* Ability to comply with study procedures and assessments

Exclusion Criteria:

* Severe psychiatric conditions requiring inpatient hospitalization (e.g., psychosis, severe major depressive episode with suicidal intent)
* Severe medical conditions requiring inpatient care (cardiovascular, renal, hematopoietic, gastrointestinal, endocrine disorders)
* Intellectual disability, illiteracy, or conditions impairing consent or questionnaire completion
* Current participation in another experimental protocol
* Active use of probiotics
* Neutropenia (<0.5 × 10^9/L)
* Leukocytosis (>30 × 10^9/L)
* Fever > 38°C
* Radiological evidence of toxic megacolon or intestinal perforation
* Presence of colostomy
* Severe comorbidity limiting 30-day survival
* Active or past malignancy requiring chemotherapy
* Corticosteroid therapy within the past 6 months
* HIV infection

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2026-11-12 (Estimated); Study Completion 2028-11-12 (Estimated)

PRIMARY OUTCOMES:
Weight | Baseline and 3 months
  Body weight measured in kilograms using a calibrated scale.
Body Mass Index (BMI) | Baseline and 3 months
  BMI calculated as weight (kg) divided by height (m²). Unit of Measure: kg/m²
Gut Microbiota Composition | Baseline and 3 months
  Assessment of the relative abundance of bacterial taxa through sequencing at baseline and 3 months. Changes over time will be evaluated to identify shifts in microbial composition and potential alterations in gut balance relevant to anorexia nervosa.
Short-Chain Fatty Acids (SCFAs) | Baseline and 3 months
  Measurement of SCFA concentrations (e.g., butyrate, acetate, propionate) at baseline and 3 months. Changes in SCFA levels will be used to evaluate alterations in gut microbial metabolic activity over time.

SECONDARY OUTCOMES:
Eating disorder psychopatology - Eating Disorder Examination Questionnaire 6.0 (EDE-Q 6.0; Calugi et al., 2015) | Baseline and 3 months
  The EDE-Q measures eating-disorder psychopathology across four subscales: Restraint, Eating Concern, Shape Concern, and Weight Concern. Items are scored from 0 to 6. The Global Score is the mean of the four subscales. Higher scores indicate more severe eating-disorder symptoms. Unit of Measure: Units on a scale.
Eating disorder psychopathology - Eating Disorder Inventory - 3 (EDI-3; Clausen et al., 2011) | Baseline and 3 months
  The EDI-3 evaluates psychological traits associated with eating disorders. It includes subscales such as Drive for Thinness, Bulimia, Body Dissatisfaction, Low Self-Esteem, Emotional Dysregulation, Interoceptive Deficits, Perfectionism, Asceticism, and others. Items are typically scored on 0-4 Likert scales. Higher scores indicate greater psychological dysfunction relevant to EDs. Unit of Measure: Units on a scale.
General psychopathology - Brief Symptom Inventory (BSI); Derogatis & Melisaratos, 1983) | Baseline and 3 months
  The BSI assesses general psychopathology. It includes the following subscales: Somatization, Obsessive-Compulsive Symptoms, Interpersonal Sensitivity, Depression, Anxiety, Hostility, Phobic Anxiety, Paranoid Ideation, and Psychoticism. Items are rated on a 0-4 scale. Higher scores indicate greater overall psychopathology. Unit of Measure: Units on a scale.
Childhood maltreatment - Childhood Trauma Questionnaire - Short Form (CTQ-SF; Bernstein et al., 2003) | Baseline
  The CTQ-SF assesses exposure to childhood maltreatment. It includes five subscales: Emotional Abuse, Physical Abuse, Sexual Abuse, Emotional Neglect, and Physical Neglect. Subscale scores range from 5 to 25; the total score ranges from 25 to 125. Higher scores indicate more severe childhood maltreatment. Unit of Measure: Units on a scale.
Emotional dysregulation - Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004) | Baseline and 3 months
  The DERS measures emotion-regulation difficulties. It includes six subscales: Nonacceptance, Goals, Impulse, Awareness, Strategies, and Clarity. Total scores range from 36 to 180. Higher scores indicate greater difficulties in emotion regulation. Unit of Measure: Units on a scale

OTHER OUTCOMES:
Inflammatory Biomarkers (pg/mL) | Baseline and 3 months
  Blood-based inflammatory markers measured in pg/mL (e.g., IL-6, TNF-α). Higher values indicate increased inflammatory activation.
C-Reactive Protein (CRP) | Baseline and 3 months
  CRP is a blood marker of systemic inflammation measured in mg/L. Higher levels indicate greater inflammatory activation.
Metabolic Biomarkers (mg/dL) | Baseline and 3 months
  Metabolic markers measured in mg/dL, including glucose and lipid profile components. Variations may reflect changes in metabolic functioning and nutritional status.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Castellini, Medical Degree, Principal Investigator — Department of Health Sciences, University of Florence, Florence, Italy
Locations (1):
- SODc Psichiatria, Azienda Ospedaliero-Universitaria Careggi, Florence, FI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quagebeur R, Dalile B, Raes J, Van Oudenhove L, Verbeke K, Vrieze E. The role of short-chain fatty acids (SCFAs) in regulating stress responses, eating behavior, and nutritional state in anorexia nervosa: protocol for a randomized controlled trial. J Eat Disord. 2023 Oct 26;11(1):191. doi: 10.1186/s40337-023-00917-6. PMID 37884972
- [Background] Mack I, Cuntz U, Gramer C, Niedermaier S, Pohl C, Schwiertz A, Zimmermann K, Zipfel S, Enck P, Penders J. Weight gain in anorexia nervosa does not ameliorate the faecal microbiota, branched chain fatty acid profiles, and gastrointestinal complaints. Sci Rep. 2016 May 27;6:26752. doi: 10.1038/srep26752. PMID 27229737
- [Background] Hata T, Miyata N, Takakura S, Yoshihara K, Asano Y, Kimura-Todani T, Yamashita M, Zhang XT, Watanabe N, Mikami K, Koga Y, Sudo N. The Gut Microbiome Derived From Anorexia Nervosa Patients Impairs Weight Gain and Behavioral Performance in Female Mice. Endocrinology. 2019 Oct 1;160(10):2441-2452. doi: 10.1210/en.2019-00408. PMID 31504398
- [Result] Facchin S, Vitulo N, Calgaro M, Buda A, Romualdi C, Pohl D, Perini B, Lorenzon G, Marinelli C, D'Inca R, Sturniolo GC, Savarino EV. Microbiota changes induced by microencapsulated sodium butyrate in patients with inflammatory bowel disease. Neurogastroenterol Motil. 2020 Oct;32(10):e13914. doi: 10.1111/nmo.13914. Epub 2020 May 31. PMID 32476236
- [Result] Castellini G, Cassioli E, Vitali F, Rossi E, Dani C, Melani G, Flaccomio D, D'Andria M, Mejia Monroy M, Galli A, Cavalieri D, Ricca V, Bartolucci GL, De Filippo C. Gut microbiota metabolites mediate the interplay between childhood maltreatment and psychopathology in patients with eating disorders. Sci Rep. 2023 Jul 20;13(1):11753. doi: 10.1038/s41598-023-38665-x. PMID 37474544